CLINICAL TRIAL: NCT06495112
Title: Comparison Between Lathe Cut Versus Cast Molding Soft Contact Lens Technique on Ocular Surface Integrity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/730
Record Dates: First submitted 2024-06-26; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Ocular Surface Disease
MeSH Terms: interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft contact lens with lathe cut technique Lathe (Other)
  Interventions: Other: Soft contact lens with lathe cut technique Lathe
- Soft contact lens with cast molding technique (Experimental)
  Interventions: Diagnostic Test: Soft contact lens with cast molding technique

INTERVENTIONS:
Other: Soft contact lens with lathe cut technique Lathe — athe cut technique Lathe cutting involves shaping a solid block of lens material into the desired form using precision machinery. This method allows for customized lens designs but may result in a less smooth surface compared to cast molding. Cast molding, on the other hand, uses a liquid monomer that is cured in a mold to form the lens. This technique typically results in a smoother and more uniform lens surface.
  Arms: Soft contact lens with lathe cut technique Lathe
Diagnostic Test: Soft contact lens with cast molding technique — Participants in this arm would receive Cast molding soft contact lenses and would wear them according to the study protocol, also likely for a specified duration.The cast molding technique for soft contact lenses involves creating lenses by polymerizing a liquid monomer mixture within a mold that forms the desired lens shape. Here's a brief overview of the steps involved in the cast molding process
  Arms: Soft contact lens with cast molding technique

SUMMARY:
"Comparison between Lathe Cut versus Cast Molding Soft Contact Lens Technique on Ocular Surface Integrity" investigates the impact of two different manufacturing methods on the health and integrity of the ocular surface.

DETAILED DESCRIPTION:
The study aims to determine which technique, lathe cutting or cast molding, produces soft contact lenses that are more biocompatible and less likely to cause adverse effects on the eye. The findings from our research could have significant implications for contact lens wearers and manufacturers, guiding the production of lenses that promote better ocular health and enhance wearer comfort. Ultimately, this research contributes valuable knowledge to optometry and ocular surface disease management.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have never used contact lenses
* Age of participants would be 15 to 35 years
* Patients free of any ocular pathology

Exclusion Criteria:

* Patients having astigmatism of more than 0.75DC
* Subjects with a previous history of ocular surgery, eye pathology, or systemic disease.
* Patients with abysmal compliance.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Corneal epithelial integrity | 12 Months
  This involves assessing the health and integrity of the outermost layer of the cornea, which can be done through optical coherence tomography (OCT)
Ocular surface symptoms | 12 months
  Utilizing standardized questionnaires or scales to assess symptoms such as dryness, discomfort, or irritation experienced by the subjects wearing the different types of soft contact lenses.

CONTACTS AND LOCATIONS:
Locations (1):
- The Keratoconus center, Eye 2 Eye Optometrists, 13 D valencia housing society, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No